CLINICAL TRIAL: NCT01432535
Title: A Single Dose Study to Assess Pharmacokinetics of SCH 54031 in Patients With Renal Impairment (P05655)
Brief Title: Pharmacokinetics of Peginterferon Alfa-2b in Participants With Moderate and Severe Renal Impairment (P05655)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05655; MK-4031-350 (Other: Merck protocol number)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Participants (Active Comparator): Participants with normal renal function defined as having a creatinine clearance test value of ≥80 mL/min/1.73 m^2. Participants receive a single subcutaneous dose of PegIFN-2b, 4.5 μg/kg.
  Interventions: Drug: PegIFN-2b (Sylatron®)
- Participants with Moderate Renal Impairment (Experimental): Participants with moderate renal impairment defined as having a creatinine clearance test value of 30-50 mL/min/1.73 m^2. Participants receive a single subcutaneous dose of PegIFN-2b, 4.5 μg/kg.
  Interventions: Drug: PegIFN-2b (Sylatron®)
- Participants with Severe Renal Impairment (Experimental): Participants with severe renal impairment defined as having a creatinine clearance test value of <30 mL/min/1.73 m^2 or end stage renal disease on hemodialysis. Participants receive a single subcutaneous dose of PegIFN-2b, 4.5 μg/kg.
  Interventions: Drug: PegIFN-2b (Sylatron®)

INTERVENTIONS:
Drug: PegIFN-2b (Sylatron®) — Single 4.5 μg/kg dose
  Other Names: PegIntron®; Peginterferon alfa-2b; SCH 054031; MK-4031

SUMMARY:
This study will compare the pharmacokinetics of a single dose of peginterferon alfa-2b (Sylatron®) in healthy participants to that in participants with moderate to severe impairment of kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 19 to 40 kg/m^2, inclusive
* Moderate renal impairment and severe renal impairment and/or end-stage renal disease (ESRD) who may require hemodialysis and normal renal function
* Free of any clinically significant disease (except those related to renal disease and comorbid conditions) that requires a physician's care and would interfere with the study
* Females of reproductive potential must have used a medically accepted method of contraception for three months prior to screening and must agree to use an accepted contraceptive method during and for two months following the study
* Males must agree to use a medically accepted method of contraception during the trial and for 3 months after the study

Exclusion Criteria:

* Pregnant, intend to become pregnant, or breastfeeding
* Surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug
* History of any infectious disease within 4 weeks prior to study drug administration that affects ability to participate in the study
* Positive for hepatitis B surface antigen, and/or for human immunodeficiency virus (HIV) antibodies. Healthy participants positive for hepatitis C antibodies
* Previously received PegIntron®, Sylatron®, and/or Pegasys
* More than 10 cigarettes or equivalent tobacco use per day
* History of malignancy
* Hypothyroidism or hyperthyroidism
* History of depression requiring treatment with psychotherapy or medication
* History of suicidality or at risk of self-harm or harm to others
* History of autoimmune disorder requiring medical therapy
* Immune mediated renal insufficiency
* Removal of a kidney (healthy participants) or functioning renal transplant (participants with renal impairment)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: Participants with normal renal function, defined as having a creatinine clearance test value of ≥80 mL/min/1.73 m^2. Participants receive a single subcutaneous dose of PegIFN-2b, 4.5 μg/kg.
Period: Overall Study
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Started | 12 | 7 (One participant later determined ineligible is not included in baseline/efficacy analyses.) | 6
Completed | 12 | 7 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment | Total
Number analyzed (Participants) | 12 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.33 (9.63) | 64.00 (6.23) | 52.67 (12.74) | 57.83 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 11 | 6 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞)
Description: AUC0-∞ is a measure of the mean concentration levels of drug in the plasma after the dose.
Time Frame: From hour 0 (pre-dose) to 288 hours post-dose
Population: All treated participants with the exception of 1 moderate renal impairment participant found to be ineligible for this arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Number analyzed (Participants) | 12 | 6 | 6
pg*hr/mL | 305315.22 [175840.19 to 530125.58] | 435500.38 [248562.28 to 763030.40] | 658413.69 [395164.74 to 10907032.58]

2. Primary Outcome: AUC From Time 0 to the Last Measurable Sample (AUC0-last)
Description: AUC0-last is a measure of the total amount of drug in the plasma from the dose to the last measurable sample.
Time Frame: From hour 0 (pre-dose) up to 288 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Number analyzed (Participants) | 12 | 6 | 6
pg*hr/mL | 286946.43 [164687.09 to 499967.87] | 408889.84 [232550.52 to 718944.43] | 598863.88 [358269.15 to 1001029.37]

3. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: From hour 0 (pre-dose) to 288 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Number analyzed (Participants) | 12 | 6 | 6
pg/mL | 2547.85 [1115.61 to 5818.84] | 3210.16 [1386.73 to 7431.24] | 3551.03 [1653.85 to 7624.49]

4. Primary Outcome: Time to Maximum Observed Serum Concentration (Tmax)
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose.
Time Frame: From hour 0 (pre-dose) up to 288 hours post-dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Number analyzed (Participants) | 12 | 6 | 6
hours | 12.0 [9.0 to 72.0] | 12.0 [12.0 to 72.0] | 60.0 [24.0 to 96.3]

5. Primary Outcome: Apparent Terminal Half-life (T1/2)
Description: T1/2 is the time required for a given drug concentration in the plasma to decrease by 50%.
Time Frame: From hour 0 (pre-dose) up to 288 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Number analyzed (Participants) | 12 | 6 | 6
Hours | 41.9 (31.9) [9.00 to 72.00] | 50.7 (12.7) [12.00 to 72.00] | 58.1 (17.2) [24.00 to 96.30]

6. Primary Outcome: Apparent Total Body Clearance (CL/F)
Description: CL/F is a calculation of the rate at which a drug is removed from the body via renal, hepatic and other clearance pathways, expressed as volume (milliliters) per unit of time (minutes).
Time Frame: From hour 0 (pre-dose) up to 288 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: mL/min
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Number analyzed (Participants) | 12 | 6 | 6
mL/min | 18.5 [10.42 to 32.85] | 12.72 [7.10 to 22.81] | 8.02 [4.71 to 13.64]

7. Primary Outcome: Apparent Volume of Distribution (Vd/F)
Description: Vd/F is defined as the distribution of a medication between the plasma and the rest of the body after the dose. It is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of the drug.
Time Frame: From hour 0 (pre-dose) up to 288 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Number analyzed (Participants) | 12 | 6 | 6
Liters | 90.63 [41.76 to 196.69] | 72.26 [32.88 to 158.82] | 55.90 [27.30 to 114.49]

ADVERSE EVENTS:
Description: One participant enrolled on the moderate renal impairment arm was later determined to be ineligible for this study arm; this participant is included in the safety analysis.
Arm/Group | Healthy Participants | Participants With Moderate Renal Impairment | Participants With Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7 | 1/6
Other Adverse Events (participants affected / at risk) | 12/12 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=12) | Participants With Moderate Renal Impairment (N=7) | Participants With Severe Renal Impairment (N=6)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=12) | Participants With Moderate Renal Impairment (N=7) | Participants With Severe Renal Impairment (N=6)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (2)
Chills (General disorders) | 9 (9) | 5 (5) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 4 (4) | 1 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 9 (9) | 6 (7) | 4 (5)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lymph node palpable (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 8 (10) | 4 (4) | 3 (3)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the Sponsor. The Investigator further agrees to provide review copies of abstracts or manuscripts for publication that report any results of the trial to the Sponsor 45 days prior to submission for publication or presentation. The Sponsor shall have the right to review and comment.